CLINICAL TRIAL: NCT00322985
Title: A Phase II Clinical Trial of Lenalidomide for T-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Celgene Corporation (Industry); Alberta Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22409
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: T-cell Lymphoma
Keywords: T-cell lymphoma; lenalidomide
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lenalidomide — 25 mg/day, orally for 21 days with 7 days rest (28 day cycle). Dosing will be in the morning at approximately the same time each day.

SUMMARY:
T-cell Non-Hodgkin's lymphomas are a group of cancers that are usually treated with chemotherapy, radiation therapy, or occasionally surgery. T-cell lymphomas are relatively uncommon and therefore not well studied. Treatment approaches are patterned after the more common B-cell lymphomas. T-cell lymphomas are more likely to relapse following standard therapy than are B-cell lymphomas. New therapies are needed for T-cell lymphomas. In this study, we will administer the drug called lenalidomide as a pill to patients with T-cell lymphoma. The goals are to determine if the drug can induce regression of the cancer, and to determine if the treatment is well tolerated in this patient group. This study will take place at six cancer centres across Canada.

DETAILED DESCRIPTION:
Background: T-cell lymphomas comprise 10-15% of all non-Hodgkin's lymphomas and include a variety of histological subtypes. These diseases have variable clinical behaviour, response to therapy, and long-term outcomes. In general, T-cell lymphomas are characterized by inferior response to therapy and prognosis compared to the more common B-cell lymphomas. Because T-cell lymphomas are uncommon, they are not generally well studied and current treatment approaches are borrowed from established protocols for B-cell lymphoma. New therapies are needed for T-cell lymphoma, and should be studied separately for their effectiveness in T-cell lymphoma.

Lenalidomide (CC-5013, Revlimid; Celgene Corporation) is an oral thalidomide analogue with anti-cancer activity. Lenalidomide is generally well tolerated, with rash, myelosuppression and venous thrombosis being the most notable and common potential side effects. Lenalidomide has demonstrated impressive anti-cancer activity against mycosis fungoides (cutaneous T-cell lymphoma), multiple myeloma, chronic lymphocytic leukemia and myelodysplasia. The drug is currently under review by Health Canada as a potential new standard therapy for multiple myeloma. We are encouraged by the efficacy and tolerability of lenalidomide in patients with related diseases, to study its role in the treatment of T-cell lymphomas other than mycosis fungoides.

Primary Objective: To determine the overall response rate to single agent lenalidomide at standard doses (25 mg po daily for 21 days of a 28-day cycle), as a treatment for T-cell lymphoma.

Secondary Objectives: To determine the complete response rate, time to progression, overall survival and tolerability for patients with T-cell lymphoma treated with lenalidomide.

Study Design: A multi-centre, Canadian, Phase II, investigator-initiated clinical trial.

Inclusion Criteria:

" Patients with the following subtypes of T-cell lymphoma:

* Peripheral T-cell lymphoma, unspecified
* Angioimmunoblastic T-cell lymphoma
* Enteropathy-type T-cell lymphoma
* NK/T-cell lymphoma
* Hepatosplenic T-cell lymphoma
* Subcutaneous panniculitic-like T-cell lymphoma
* Anaplastic large cell lymphoma
* Lymphoblastic T-cell lymphoma " Measurable disease (See section 6.2) " WHO performance status of 0-2 " Both untreated patients with contraindications to chemotherapy, and patients with relapsed/refractory disease after at least one line of chemotherapy are allowed; no restriction on the number of prior therapies " Patients with prior radiotherapy, autologous or allogeneic stem cell transplant are allowed " Age >18 years, able to give informed consent " Acceptable hematological and biochemical parameters (see section 6.2)

Exclusion Criteria:

" Mycosis Fungoides/Sezary Syndrome " Pregnant or lactating females " Concurrent use of other anti-cancer therapies " Other serious co-morbid illness that would compromise participation in the study " Prior therapy with lenalidomide " Prior hypersensitivity to thalidomide

It is intended to enroll patients who have relapsed in spite of chemotherapy, radiotherapy and/or high dose therapy with stem cell transplant, or patients who are not eligible for these standard therapies. It would be encouraged that patients are initially treated with standard therapy if possible. However, we wish to allow untreated patients to participate because older, frail patients with disseminated T-cell lymphoma or patients with significant comorbidities may not be eligible for aggressive chemotherapy but may tolerate lenalidomide quite well. In this regard, it is left to the discretion of the investigator to determine whether or not an individual patient should be considered for enrollment on this clinical trial, or whether that patient would be better served with standard treatment approaches.

Recruitment will take place in the outpatient clinics of the Cross Cancer Institute and five other Canadian cancer clinics (Vancouver, Calgary, Winnipeg, Ottawa, Halifax). The Cross Cancer Institute will be the lead site for the trial and our team will be responsible for oversight of the trial, collation of patient case report forms, communication with Health Canada and Celgene, and data analysis. Celgene will monitor all the sites involved in the trial every 3-4 months.

Statistical Analysis will use standard methods and will include a data safety and monitoring committee (DSMB) who will perform interim safety analyses after ten and 22 patients have been enrolled on trial. An interim efficacy analysis will be performed after 22 patients have been enrolled. The trial will be stopped if fewer than 2 of the first 22 patients enrolled achieve an objective response to therapy according to standard criteria. If two or more responses occur, the trial will continue until the remaining 18 patients will be accrued in the absence of safety concerns. There are no pre-specified criteria for stopping the trial on the basis of safety concerns, but the investigators and the independent DSMB will each have the power to halt enrollment if serious safety concerns arise at any point during the trial. Patients will be required to stop the study treatment if severe adverse reactions occur, the lymphoma progresses, serious intercurrent illness interferes with treatment, suspected pregnancy occurs, or for major study protocol violations.

Sample size: For a total of 40 subjects, 22 will be accrued during stage 1 and 18 during stage 2. If 1 or fewer responses are observed during the first stage then the trial is stopped early. Given that the 'true' response probability is 5%, there is a 70% probability of ending the trial during stage 1. However, if the 'true' response probability is 20% then there is a 5% probability that the trial will be stopped in stage 1. The alpha level of the design is 0.04 and the power is 0.9. If fewer than 4 of 40 patients respond, this will be considered evidence that lenalidomide is inactive in the population studied.

ELIGIBILITY:
Inclusion Criteria:

* T-cell lymphoma (excluding mycosis fungoides)
* WHO performance status 0-2
* measurable lesions
* acceptable hematological and biochemical parameters
* previously treated OR untreated but not suitable for standard therapy

Exclusion Criteria:

* pregnant
* HIV
* viral hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
overall response rate | every 3 months
  Defined by the Cheson criteria for response in lymphoma and will be expressed as percentages

SECONDARY OUTCOMES:
complete response rate | every 3 months
  Defined by the Cheson criteria for response in lymphoma and will be expressed as percentages.
Time To Progression [TTP] | every 3 months
  Kaplan-Meier curves will be used to plot Time to Progression.
survival | every 3 months
  Kaplan-Meier curves will be used to plot survival.
safety | every 3 months
  The severity of the toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v3 whenever possible. The first interim safety analysis will be conducted by the Data Monitoring Committee after the first 10 patients have completed therapy on trial. This safety analysis will be repeated at the second interim analysis of 22 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Reiman, MD, Principal Investigator — Alberta Health services
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II, Health Services Centre, Halifax, Nova Scotia
  - Ottawa Hospital General Campus, Ottawa, Ontario

REFERENCES:
- [Derived] Toumishey E, Prasad A, Dueck G, Chua N, Finch D, Johnston J, van der Jagt R, Stewart D, White D, Belch A, Reiman T. Final report of a phase 2 clinical trial of lenalidomide monotherapy for patients with T-cell lymphoma. Cancer. 2015 Mar 1;121(5):716-23. doi: 10.1002/cncr.29103. Epub 2014 Oct 29. PMID 25355245